CLINICAL TRIAL: NCT05110781
Title: Neo-Adjuvant Atezolizumab Prior to Definitive Surgical Resection of Regionally Metastatic Head &Amp; Neck Cutaneous Squamous Cell Carcinoma With an Unknown or Historic Primary Site: A Window Trial
Brief Title: Atezolizumab Before Surgery for the Treatment of Regionally Metastatic Head and Neck Squamous Cell Cancer With an Unknown or Historic Primary Site
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Arnaud Bewley, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Arnaud Bewley, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#295; NCI-2021-10734 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#295 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2021-10-13; First posted 2021-11-08 (Actual); Results first posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced Cutaneous Squamous Cell Carcinoma of the Head and Neck; Resectable Cutaneous Squamous Cell Carcinoma of the Head and Neck; Stage III Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8
MeSH Terms: interventions — atezolizumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (atezolizumab, surgery, radiation therapy) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery. Beginning 6 weeks after surgery, patients with residual disease undergo standard of care radiation therapy and receive atezolizumab IV over 30-60 minutes on day 1. Treatment with atezolizumab repeats every 21 days for up to 15 cycles in the absence of disease progression and unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase II trial tests whether atezolizumab works to shrink tumors before surgery in patients with head and neck squamous cell cancer with an unknown or historic primary site that has spread to other places in the lymph nodes (regionally metastatic). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving atezolizumab before surgery may reduce the size of the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:I. Evaluate the rate of pathologic complete response (pCR) at the time of surgery following neo-adjuvant atezolizumab in patients with regionally metastatic head and neck cutaneous squamous cell carcinoma (HNSCCC).

SECONDARY OBJECTIVES:I. Further characterize the oncologic response to neo-adjuvant atezolizumab and adjuvant atezolizumab in combination with radiation therapy in patients with regionally metastatic HNSCCC:Ia. Determine the rate of major pathologic response (mPR) at the time of surgery.Ib. Evaluate the 2-year event free survival (EFS) after completion of adjuvant therapy.

II. Investigate the utility of conventional imaging and novel biomarkers in predicting and assessing response to neoadjuvant atezolizumab therapy.IIa. Investigate associations between pre-treatment tumor fludeoxyglucose F-18 (FDG) avidity and response to neoadjuvant immunotherapy.IIb. Evaluate the ability of fine-cut contrast enhanced computed tomography (CT) or magnetic resonance imaging (MRI) of the head and neck to assess response to neoadjuvant immunotherapy prior to surgery.IIc. Evaluate the capabilities of serial liquid biopsy analysis of tumor-associated exosomes to predict neoadjuvant immunotherapy response.

III. Evaluate the safety and tolerability of anti-PD-L1 with atezolizumab neo-adjuvant therapy in resectable regional metastatic HNCSCC.IIIa. Quantify toxicity (adverse events) determined by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.

OUTLINE:Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery. Beginning 6 weeks after surgery, patients with residual disease undergo standard of care radiation therapy and receive atezolizumab IV over 30-60 minutes on day 1. Treatment with atezolizumab repeats every 21 days for up to 15 cycles in the absence of disease progression and unacceptable toxicity.After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants with biopsy proven, surgically resectable head and neck cutaneous squamous cell carcinoma regionally metastatic to lymph nodes in the head and/or neck with a historical or unknown (but not concurrent) primary site
* Patients must be >= 18 years
* Patients with resectable regionally metastatic HNCSCC from an unknown or historical primary and no evidence of distant metastatic disease
* Full decision-making capacity and consent provided and documented
* Radiographically measurable disease per immune Response Evaluation Criteria in Solid Tumors (iRECIST)
* Surgically resectable disease per standard of care (SoC)
* For Women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods as defined below: * Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the final dose of atezolizumab * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception
* Men: abstinent or using effective contraception method
* Tumor tissue sample adequate for PD-L1 and biomarker studies
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Availability of a representative tumor specimen for exploratory biomarker research
* Life expectancy >= 2 years
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (1500/uL) without granulocyte colony-stimulating factor support (within 14 days prior to initiation of study treatment)
* Lymphocyte count >= 0.5 x 10^9/L (500/uL) (within 14 days prior to initiation of study treatment)
* Platelet count >= 50 x 10^9/L (50,000/uL) without transfusion (within 14 days prior to initiation of study treatment)
* Hemoglobin >= 80 g/L (8 g/dL) (within 14 days prior to initiation of study treatment) * Patients may be transfused to meet this criterion
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) =< 2.5 x upper limit of normal (ULN) (within 14 days prior to initiation of study treatment)
* Serum bilirubin =< 1.5 x ULN (within 14 days prior to initiation of study treatment) with the following exception: * Patients with known Gilbert disease: serum bilirubin =< 3 x ULN
* Serum creatinine =< 1.5 x ULN or creatinine clearance >= 60 mL/min (calculated using the Cockcroft-Gault formula (within 14 days prior to initiation of study treatment)
* Serum albumin >= 25 g/L (2.5 g/dL) (within 14 days prior to initiation of study treatment)
* For patients not receiving therapeutic anticoagulation: international normalized ratio (INR) or activated partial thromboplastin time (aPTT) =< 1.5 x ULN
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Negative human immunodeficiency virus (HIV) test at screening with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count >= 200, and have an undetectable viral load
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) deoxyribonucleic acid (DNA) test at screening
* The HBV DNA test will be performed only for patients who have a negative HBsAg test and a positive total HBcAb test

Exclusion Criteria:

* Distant metastatic disease
* Unresectable disease: As defined by: common or internal carotid artery encasement or involvement of the skull base involvement or pre-vertebral fascia
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) * Patients with indwelling catheters (e.g., PleurX) are allowed
* Uncontrolled (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions: * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met: ** Rash must cover < 10% of body surface area ** Disease is well controlled at baseline and requires only low-potency topical corticosteroids ** No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months * Any history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Known active tuberculosis
* Significant cardiovascular disease (such as New York Heart Association class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival [OS] rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia. Severe infection is defined as that requiring inpatient treatment of hospitalization
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment * Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 6 months after the final dose of atezolizumab
* Current treatment with anti-viral therapy for HBV. Patient on suppressive therapy should excluded
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions: * Patients who received acute, low-dose (defined as < 200 mg / day hydrocortisone or equivalent) corticosteroid treatment (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after principal investigator confirmation has been obtained * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Concurrent identifiable primary cutaneous head and neck squamous cell carcinoma tumor
* Pregnant or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2023-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bewley, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not applicable; only one participant was enrolled and the enrolled participant received study treatment.
Period: Overall Study
Arm/Group | Treatment (Atezolizumab, Surgery, Radiation Therapy)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Atezolizumab, Surgery, Radiation Therapy)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: Years] | 78 [78 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR)
Description: pCR is defined as having no residual invasive squamous cell carcinoma within the primary tumor and all resected lymph nodes as assessed by the pathologist at the time of primary resection. The rate of pCR is defined as the proportion of patients demonstrating pCR.
Time Frame: At time of surgery (up to 10 weeks from time of enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Atezolizumab, Surgery, Radiation Therapy)
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Major Pathologic Response (mPR)
Description: mPR is defined as having =< 10% residual invasive squamous cell carcinoma within the primary tumor and all resected lymph nodes as assessed by the pathologist at the time of primary resection. The rate of mPR is defined as the proportion of patients demonstrating mPR.
Time Frame: At time of surgery (up to 10 weeks from time of enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Atezolizumab, Surgery, Radiation Therapy)
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Number of Participants With Recurrence or Disease Progression
Description: A non-parametric Kaplan-Meier (KM) method will be used to estimate the 2-year EFS curve. Participants who do not experience recurrence or disease progression at the time of their last follow-up will be censored. Recurrence, all-cause death and disease-specific death will be likewise examined using the KM method to determine estimates of 2-yr disease-free survival, overall survival and disease-specific survival.
Time Frame: From randomization to the first day of radiographic evidence of recurrence or disease progression, clinical evidence of recurrence or disease progression, or death due to any cause, whichever occurs first, assessed at 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Atezolizumab, Surgery, Radiation Therapy)
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Standardized Uptake Value (SUV) of Primary Lesion Assessed at Baseline and 3 Months After Completion of Treatment
Description: FDG avidity of nodal sites will be quantified according to standardized uptake value (SUV). The SUV is the ratio of the image derived radioactivity concentration of the lesion of interest and the whole body concentration of the injected radioactivity. Standard of care staging positron emission tomography (PET)/computed tomography (CT) will be performed prior to initiation of treatment and as a post-treatment scan 3 months after completion. The association of the SUV of the regionally metastatic focus of disease to the pathologic response to neoadjuvant therapy at the time of surgery will be examined. A t-test (or nonparametric counterpart) and multiple regression will be used to compare mean SUV between patients who experience cPR to the mean SUV of those with residual disease after neoadjuvant therapy, where the latter will adjust patient characteristics and potential confounders. In addition, the mean SUV of additional sites of regionally metastatic disease will be studied.
Time Frame: At baseline and 3 months after completion of treatment
Measure: Number; unit: Ratio
Arm/Group | Treatment (Atezolizumab, Surgery, Radiation Therapy)
Number analyzed (Participants) | 1
Ratio
  Baseline SUV | 9.2
  Month 3 SUV | 2.99

5. Secondary Outcome: Number of Participants With Overall Response
Description: Measured by CT or magnetic resonance imaging (MRI) of the head and neck per immune Response Evaluation Criteria in Solid Tumors (iRECIST) criteria.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Atezolizumab, Surgery, Radiation Therapy)
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Plasma Exosome Levels
Time Frame: Up to 3 years
Population: Plasma exosome level was not measured as the study was terminated early due to low accrual and only 1 evaluable participant was enrolled.
Arm/Group | Treatment (Atezolizumab, Surgery, Radiation Therapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Adverse Events
Description: Determined by Common Terminology Criteria for Adverse Events version 5. Safety and tolerability will be assessed by clinical review of all relevant parameters including adverse events, laboratory tests, and vital signs. Descriptive statistics will be provided for adverse events.
Time Frame: From study treatment initiation through 1 year post-surgery
Measure: Number; unit: adverse events
Arm/Group | Treatment (Atezolizumab, Surgery, Radiation Therapy)
Number analyzed (Participants) | 1
adverse events | 3

ADVERSE EVENTS:
Time Frame: From study treatment initiation through 1 year post-surgery
Arm/Group | Treatment (Atezolizumab, Surgery, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Atezolizumab, Surgery, Radiation Therapy) (N=1)
Edema face (General disorders) | 1 (1)
Pain (General disorders) | 1 (1) — Intermittent sharp pain at surgical site.
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Discomfort when swallowing.

LIMITATIONS AND CAVEATS:
One participant was enrolled in study prior to termination. Enrollment in the clinical trial did not reach the target number of participants needed to achieve target power and was insufficient to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT05110781/Prot_SAP_000.pdf